CLINICAL TRIAL: NCT04559698
Title: Assessing Mental Health Providers' Clinical Knowledge and Skills Via an Online Training on LGBTQ-affirmative Cognitive-behavioral Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: David R. Kessler, M.D. '55 Fund for LGBTQ Mental Health Research at Yale (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2000028914
Record Dates: First submitted 2020-09-16; First posted 2020-09-23 (Actual); Results first posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: LGBTQ

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate training group (Experimental): Participants will take part in 11-week LGBTQ-affirmative CBT training via Zoom for 1-hour per week. The participants in the immediate training group will take part in the first 11-week course.
  Interventions: Behavioral: LGBTQ-affirmative CBT training
- waitlist control group (Experimental): Participants will take part in 11-week LGBTQ-affirmative CBT training via Zoom for 1-hour per week. The participants in the waitlist control group will take part in the second 11-week course.
  Interventions: Behavioral: LGBTQ-affirmative CBT training

INTERVENTIONS:
Behavioral: LGBTQ-affirmative CBT training — Participants will take part in 11-week LGBTQ-affirmative CBT training via Zoom for 1-hour per week.

SUMMARY:
The purpose of the proposed study is to train mental health providers (MHPs) at lesbian, gay, bisexual, transgender, and queer (LGBTQ) community centers across the United States in evidence-based, LGBTQ-affirmative cognitive-behavioral therapy (CBT).

DETAILED DESCRIPTION:
The purpose of the proposed study is to train mental health providers (MHPs) at LGBTQ community centers across the United States in evidence-based, LGBTQ-affirmative cognitive-behavioral therapy (CBT).

The primary objective of this study is to determine whether the LGBTQ-affirmative CBT training increases LGBTQ and CBT knowledge, clinical skills, and cultural humility among a sample of MHPs from LGBTQ community centers in the U.S. The proposed prospective study will follow a 2-arm waitlist randomized-controlled trial design where one group of MHPs will be randomized to receive the intervention training (i.e., the immediate training group) in LGBTQ-affirmative CBT, and the second group of MHPs will be randomized to a waitlist control group.

The proposed mixed-methods study will consist of predominantly quantitative self-report measures, as well as a qualitative self-assessment of participants' LGBTQ-affirmative CBT clinical skills. All study measures will be administered online at three time points-- baseline, 4-months post-baseline, and 8-months post-baseline (changed prior to randomization from 3-months and 6-months, respectively)-- via the secure Yale Qualtrics survey software.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* Fluent in English
* Mental health provider (including, but not limited to licensed practicing counselors, licensed clinical social workers, licensed marital and family therapists, clinical/counseling psychologists, pre-doctoral psychology interns, third-year or greater graduate practicum students/externs)
* Currently practicing in an LGBTQ community center that is coordinated by CenterLink, the coordinating hub for LGBTQ community centers in the U.S.

Exclusion Criteria:

* • Individuals unwilling or unable to give informed consent at the time of participation and/or not fitting the eligibility criteria outlined above

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06-26 (Actual); Study Completion 2021-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Pachankis, Ph.D., Principal Investigator — Associate Professor of Public Health (Social and Behavioral Sciences)
Locations (1):
- Yale LGBTQ+ Mental Health Initiative - Research Lab, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bidell, M. P. (2005). The Sexual Orientation Counselor Competency Scale: Assessing attitudes, skills, and knowledge of counselors working with lesbian, gay, and bisexual clients. Counselor Education and Supervision, 44(4), 267-279.
- [Background] Gonzalez, E., Sperandio, K. R., Mullen, P. R., & Tuazon, V. E. (2021). Development and initial testing of the Multidimensional Cultural Humility Scale. Measurement and Evaluation in Counseling and Development, 54(1), 56-70.
- [Background] Meyer IH. Prejudice, social stress, and mental health in lesbian, gay, and bisexual populations: conceptual issues and research evidence. Psychol Bull. 2003 Sep;129(5):674-697. doi: 10.1037/0033-2909.129.5.674. PMID 12956539
- [Background] Pachankis JE, McConocha EM, Clark KA, Wang K, Behari K, Fetzner BK, Brisbin CD, Scheer JR, Lehavot K. A transdiagnostic minority stress intervention for gender diverse sexual minority women's depression, anxiety, and unhealthy alcohol use: A randomized controlled trial. J Consult Clin Psychol. 2020 Jul;88(7):613-630. doi: 10.1037/ccp0000508. Epub 2020 May 21. PMID 32437174
- [Background] Myles, P. J., & Milne, D. L. (2004). Outcome evaluation of a brief shared learning programme in cognitive behavioural therapy. Behavioural and Cognitive Psychotherapy, 32(2), 177-188.
- [Background] White Hughto JM, Clark KA, Altice FL, Reisner SL, Kershaw TS, Pachankis JE. Improving correctional healthcare providers' ability to care for transgender patients: Development and evaluation of a theory-driven cultural and clinical competence intervention. Soc Sci Med. 2017 Dec;195:159-169. doi: 10.1016/j.socscimed.2017.10.004. Epub 2017 Oct 30. PMID 29096945
- [Background] Lelutiu-Weinberger C, Pachankis JE. Acceptability and Preliminary Efficacy of a Lesbian, Gay, Bisexual, and Transgender-Affirmative Mental Health Practice Training in a Highly Stigmatizing National Context. LGBT Health. 2017 Oct;4(5):360-370. doi: 10.1089/lgbt.2016.0194. Epub 2017 Sep 11. PMID 28891750
- [Background] Rousmaniere, T. (2017). Deliberate practice for psychotherapists: A guide to improving clinical effectiveness. Routledge/Taylor & Francis Group.
- [Derived] Pachankis JE, Soulliard ZA, Seager van Dyk I, Layland EK, Clark KA, Levine DS, Jackson SD. Training in LGBTQ-affirmative cognitive behavioral therapy: A randomized controlled trial across LGBTQ community centers. J Consult Clin Psychol. 2022 Jul;90(7):582-599. doi: 10.1037/ccp0000745. PMID 35901370

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted through an online flyer emailed to listservs of mental health providers at CenterLink LGBTQ community centers. An informal webinar was also held in October 2020 for mental health providers at CenterLink LGBTQ community centers to learn more about the study.
Period: Overall Study
Arm/Group | Immediate Training Group | Waitlist Control Group
Started | 61 | 60
Four-month Pre-intervention | 0 (Participants in this arm started training immediately after randomization, and therefore, did not have a four-month waiting period prior to receiving the training.) | 60
Immediate Pre-intervention | 61 | 55
Immediate Post-intervention | 52 | 44
Four-month Post-intervention | 47 | 0 (Participants in this arm started training four months after randomization (waitlist) and therefore, were not assessed at the four-month follow-up time point due to completion of the study.)
Completed | 47 | 44
Not Completed | 14 | 16
Not completed — Lost to Follow-up | 14 | 15
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Training Group | Waitlist Control Group | Total
Number analyzed (Participants) | 61 | 60 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.74 (11.36) | 35.72 (9.33) | 37.74 (10.55)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Participants were allowed to select more than one option for gender identity, leading to n > 121 for this measure.
  Participants
    Gender Identity : Cisgender Man | 14 | 11 | 25
    Gender Identity : Cisgender Woman | 29 | 37 | 66
    Gender Identity : Transgender Man | 6 | 0 | 6
    Gender Identity : Transgender Woman | 1 | 1 | 2
    Gender Identity : Gender Non-Binary | 4 | 8 | 12
    Gender Identity : Gender Non-Conforming | 1 | 2 | 3
    Gender Identity : Genderqueer | 6 | 1 | 7
    Gender Identity : Other | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 9 | 24
  Not Hispanic or Latino | 46 | 51 | 97
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 8 | 13
  White | 43 | 38 | 81
  More than one race | 11 | 11 | 22
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 60 | 59 | 119
  Canada | 1 | 0 | 1
  Uganda | 0 | 1 | 1
Sexual Orientation [Count of Participants; unit: Participants]
  Asexual | 1 | 1 | 2
  Bisexual | 6 | 7 | 13
  Gay | 13 | 9 | 22
  Heterosexual/Straight | 14 | 14 | 28
  Lesbian | 9 | 9 | 18
  Pansexual | 7 | 6 | 13
  Queer | 11 | 13 | 24
  Other | 0 | 1 | 1
Education Degree [Count of Participants; unit: Participants]
  High School/GED or Associate's Degree | 2 | 0 | 2
  Bachelor's Degree | 6 | 14 | 20
  Master's Degree | 50 | 45 | 95
  Doctoral Degree | 3 | 1 | 4
Employment Status [Count of Participants; unit: Participants]
  Full-Time (40 Hours Per Week) | 37 | 29 | 66
  Part-Time (Less Than 40 Hours Per Week) | 19 | 12 | 31
  Practicum Student/Intern | 3 | 13 | 16
  Other | 2 | 6 | 8
Theoretical Orientation [Count of Participants; unit: Participants]
  Cognitive Behavioral (CBT) | 10 | 17 | 27
  Existential | 0 | 1 | 1
  Humanistic/Person-Centered | 15 | 14 | 29
  Psychodynamic/Psychoanalytic | 2 | 3 | 5
  Solution-Focused | 9 | 4 | 13
  Third-Wave CBT | 1 | 0 | 1
  Eclectic or Integrative | 23 | 21 | 44
  Missing | 1 | 0 | 1
Primary Mode of Psychotherapy [Count of Participants; unit: Participants]
  Individual Therapy | 52 | 46 | 98
  Family Therapy | 1 | 0 | 1
  Group Therapy | 7 | 9 | 16
  Other | 1 | 5 | 6
Age of Clients [Count of Participants; unit: Participants]
  <5-12 | 2 | 2 | 4
  13-17 | 5 | 7 | 12
  18-30 | 29 | 29 | 58
  31-50 | 23 | 19 | 42
  51-65+ | 2 | 3 | 5
Number of Years Working in Mental Health [Mean (Standard Deviation); unit: years] | 6.85 (7.42) | 5.40 (6.77) | 6.13 (7.11)
Number of Years Working with LGBTQ Clients [Mean (Standard Deviation); unit: years] | 4.33 (5.37) | 2.82 (2.95) | 3.58 (4.39)

OUTCOME MEASURES:

1. Primary Outcome: Familiarity With LGBTQ-Affirmative CBT Skills
Description: Familiarity with LGBTQ-affirmative CBT skills will be measured using a self-developed questionnaire by the researchers for the purpose of this study. This questionnaire consists of 7 items rated on a 5-point Likert scale for each item. An overall score of 35 (sum of all items) would be the highest possible score on the questionnaire and would indicate a high level of familiarity with LGBTQ-affirmative CBT skills.
Time Frame: Four-month Pre-intervention, Immediate Pre-intervention, Immediate Post-intervention, Four-month Post-intervention
Population: Participants in the Immediate training group started training immediately after randomization, and therefore, have no data for the four-month waiting period prior to receiving the intervention. Participants in the Waitlist control group started training four months after randomization and therefore, were not assessed at the four-month follow-up time point due to completion of the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Immediate Training Group | Waitlist Control Group
Number analyzed (Participants) | 61 | 60
score on a scale
  Four-month Pre-intervention: number analyzed (Participants) | 0 | 60
  Four-month Pre-intervention |  | 19.00 (0.66)
  Immediate Pre-intervention: number analyzed (Participants) | 61 | 55
  Immediate Pre-intervention | 18.30 (0.76) | 19.70 (0.76)
  Immediate Post-intervention: number analyzed (Participants) | 52 | 44
  Immediate Post-intervention | 24.34 (0.66) | 25.46 (0.79)
  Four-month Post-intervention: number analyzed (Participants) | 47 | 0
  Four-month Post-intervention | 25.57 (0.66) |

2. Primary Outcome: Use of LGBTQ-Affirmative CBT Skills
Description: Use LGBTQ-affirmative CBT skills will be measured using a self-developed questionnaire by the researchers for the purpose of this study. This questionnaire consists of 7 items rated on a 5-point Likert scale for each item. An overall score of 35 (sum of all items) would be the highest possible score on the questionnaire and would indicate a high level of use of LGBTQ-affirmative CBT skills.
Time Frame: Four-month Pre-intervention, Immediate Pre-intervention, Immediate Post-intervention, Four-month Post-intervention
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Immediate Training Group | Waitlist Control Group
Number analyzed (Participants) | 61 | 60
score on a scale
  Four-month Pre-intervention: number analyzed (Participants) | 0 | 60
  Four-month Pre-intervention |  | 17.53 (0.66)
  Immediate Pre-intervention: number analyzed (Participants) | 61 | 55
  Immediate Pre-intervention | 16.77 (0.67) | 18.46 (0.77)
  Immediate Post-intervention: number analyzed (Participants) | 52 | 44
  Immediate Post-intervention | 22.93 (0.72) | 23.61 (0.77)
  Four-month Post-intervention: number analyzed (Participants) | 47 | 0
  Four-month Post-intervention | 24.02 (0.69) |

3. Secondary Outcome: Self-Reported LGBTQ Clinical Skills Competency
Description: Competency in LGBTQ clinical skills will be measured using the Sexual Orientation Counselor Competency Scale (SOCCS) - Clinical Skills subscale. This subscale consists of 11-items from a psychometrically validated measure, based on a 7-point Likert scale assessing the extent to which respondents endorse clinical competence as related to their skills in working with clients of diverse sexual identities. For the present study, items have been adapted to specifically assess competence in clinical skills based on an LGBTQ-affirmative CBT framework. An overall score of 7 (arithmetic mean of all 11 items) would be the highest possible score and would indicate a high level of competence in LGBTQ clinical skills.
Time Frame: Four-month Pre-intervention, Immediate Pre-intervention, Immediate Post-intervention, Four-month Post-intervention
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Immediate Training Group | Waitlist Control Group
Number analyzed (Participants) | 61 | 60
score on a scale
  Four-month Pre-intervention: number analyzed (Participants) | 0 | 60
  Four-month Pre-intervention |  | 3.30 (0.19)
  Immediate Pre-intervention: number analyzed (Participants) | 61 | 55
  Immediate Pre-intervention | 3.31 (0.17) | 3.14 (0.18)
  Immediate Post-intervention: number analyzed (Participants) | 52 | 44
  Immediate Post-intervention | 5.05 (0.15) | 5.03 (0.19)
  Four-month Post-intervention: number analyzed (Participants) | 47 | 0
  Four-month Post-intervention | 5.33 (0.13) |

4. Secondary Outcome: Applied LGBTQ Clinical Skills Competency
Description: Competency in LGBTQ clinical skills will be measured by asking participants to provide responses to videos of fictional LGBTQ clients. Participants will watch 2 brief video clips (90 seconds each) of fictional clients presenting concerns they would like to address in psychotherapy. Participants will then be asked to write a brief paragraph describing what clinical approaches they would use in clinical treatment in order to address the challenges discussed by the fictional client. These written responses will be rated based on 22 items on a 2-point scale of 0 (did not mention at all), 1 (briefly discussed), and 2 (discussed in detail) to determine participants' LGBTQ-affirmative and general CBT skills. Items coded related to LGBTQ-affirmative CBT skills will not be double coded in the comparable items related to general CBT skills. Average scores will be taken such that 2 would be the highest possible score and would indicate a high level of competence in LGBTQ clinical skills.
Time Frame: Four-month Pre-intervention, Immediate Pre-intervention, Immediate Post-intervention, Four-month Post-intervention
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Immediate Training Group | Waitlist Control Group
Number analyzed (Participants) | 61 | 60
score on a scale
  Four-month Pre-intervention: number analyzed (Participants) | 0 | 60
  Four-month Pre-intervention |  | 0.12 (0.02)
  Immediate Pre-intervention: number analyzed (Participants) | 61 | 55
  Immediate Pre-intervention | 0.11 (0.02) | 0.14 (0.02)
  Immediate Post-intervention: number analyzed (Participants) | 52 | 44
  Immediate Post-intervention | 0.24 (0.03) | 0.31 (0.03)
  Four-month Post-intervention: number analyzed (Participants) | 47 | 0
  Four-month Post-intervention | 0.22 (0.03) |

5. Secondary Outcome: Applied CBT Clinical Skills Competency
Description: Competency in general CBT clinical skills will be measured by asking participants to provide responses to videos of fictional LGBTQ clients. Participants will watch 2 brief video clips (90 seconds each) of fictional clients presenting concerns they would like to address in psychotherapy. Participants will then be asked to write a brief paragraph describing what clinical approaches they would use in clinical treatment in order to address the challenges discussed by the fictional client. These written responses will be rated based on 22 items on a 2-point scale of 0 (did not mention at all), 1 (briefly discussed), and 2 (discussed in detail) to determine participants' LGBTQ-affirmative and general CBT skills. Items coded related to LGBTQ-affirmative CBT skills will not be double coded in the comparable items related to general CBT skills. Average scores will be taken such that 2 would be the highest possible score and would indicate a high level of competence in CBT clinical skills.
Time Frame: Four-month Pre-intervention, Immediate Pre-intervention, Immediate Post-intervention, Four-month Post-intervention
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Immediate Training Group | Waitlist Control Group
Number analyzed (Participants) | 61 | 60
units on a scale
  Four-month Pre-intervention: number analyzed (Participants) | 0 | 60
  Four-month Pre-intervention |  | 0.12 (0.01)
  Immediate Pre-intervention: number analyzed (Participants) | 61 | 55
  Immediate Pre-intervention | 0.10 (0.01) | 0.12 (0.01)
  Immediate Post-intervention: number analyzed (Participants) | 52 | 44
  Immediate Post-intervention | 0.17 (0.03) | 0.11 (0.02)
  Four-month Post-intervention: number analyzed (Participants) | 47 | 0
  Four-month Post-intervention | 0.14 (0.02) |

6. Secondary Outcome: LGBTQ Cultural Humility
Description: LGBTQ cultural humility will be measured using the Multidimensional Cultural Humility Scale (MCHS). This questionnaire is a 15-item self-report psychometrically validated measure assessing the extent to which respondents endorse an ability to maintain an other-oriented, interpersonal stance in relation to cultural identities most salient to clients. For the present study, items were adapted to specifically assess cultural humility as related to working with LGBTQ clients. An overall score of 90 (sum of all items) would be the highest possible score on the questionnaire and would indicate a high level of LGBTQ cultural humility.
Time Frame: Four-month Pre-intervention, Immediate Pre-intervention, Immediate Post-intervention, Four-month Post-intervention
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Immediate Training Group | Waitlist Control Group
Number analyzed (Participants) | 61 | 60
score on a scale
  Four-month pre-intervention: number analyzed (Participants) | 0 | 60
  Four-month pre-intervention |  | 75.28 (0.83)
  Immediate pre-intervention: number analyzed (Participants) | 61 | 55
  Immediate pre-intervention | 76.48 (0.90) | 75.76 (1.03)
  Immediate post-intervention: number analyzed (Participants) | 52 | 44
  Immediate post-intervention | 77.34 (0.88) | 77.27 (1.27)
  Four-month Post-intervention: number analyzed (Participants) | 47 | 0
  Four-month Post-intervention | 78.55 (0.74) |

7. Secondary Outcome: Content Knowledge of Minority Stress
Description: Content knowledge of minority stress will be measured using a self-developed, 10-item multiple-choice measure by the researchers for the purpose of this study and based on past minority stress research. An overall score of 10 (i.e., answering all 10-items correctly) would be the highest possible score on the measure and would indicate a high level of content knowledge of minority stress.
Time Frame: Four-month Pre-intervention, Immediate Pre-intervention, Immediate Post-intervention, Four-month Post-Intervention
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Immediate Training Group | Waitlist Control Group
Number analyzed (Participants) | 61 | 60
score on a scale
  Four-month Pre-intervention: number analyzed (Participants) | 0 | 60
  Four-month Pre-intervention |  | 7.15 (0.19)
  Immediate Pre-intervention: number analyzed (Participants) | 61 | 55
  Immediate Pre-intervention | 7.02 (0.19) | 7.04 (0.26)
  Immediate Post-intervention: number analyzed (Participants) | 52 | 44
  Immediate Post-intervention | 8.05 (0.21) | 7.63 (0.34)
  Four-month Post-intervention: number analyzed (Participants) | 47 | 0
  Four-month Post-intervention | 7.82 (0.24) |

8. Secondary Outcome: Content Knowledge of CBT/LGBTQ-Affirmative CBT
Description: Content knowledge of CBT/LGBTQ-affirmative CBT will be measured using a self-developed, 10-item multiple-choice measure by the researchers for the purpose of this study based on past interventional studies of LGBTQ-affirmative CBT. An overall score of 10 (i.e., answering all 10-items correctly) would be the highest possible score on the measure and would indicate a high level of content knowledge of CBT/LGBTQ-affirmative CBT.
Time Frame: Four-month Pre-intervention, Immediate Pre-intervention, Immediate Post-intervention, Four-month Post-intervention
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Immediate Training Group | Waitlist Control Group
Number analyzed (Participants) | 61 | 60
score on a scale
  Four-month Pre-intervention: number analyzed (Participants) | 0 | 60
  Four-month Pre-intervention |  | 5.48 (0.21)
  Immediate Pre-intervention: number analyzed (Participants) | 61 | 55
  Immediate Pre-intervention | 5.36 (0.24) | 5.46 (0.26)
  Immediate Post-intervention: number analyzed (Participants) | 52 | 44
  Immediate Post-intervention | 6.77 (0.30) | 6.80 (0.32)
  Four-month Post-intervention: number analyzed (Participants) | 47 | 0
  Four-month Post-intervention | 6.48 (0.28) |

9. Secondary Outcome: Acceptability of LGBTQ-affirmative CBT Training
Description: Acceptability of LGBTQ-affirmative CBT will measured using a self-developed questionnaire by the researchers based on past research on training acceptability. Participants will be asked to report how many of the 11 training sessions they attended. Participants will then be asked 2 qualitative questions in regard to which of the 11 training sessions they found most and least helpful. Participants will also be asked 7 questions based on a 5-point Likert scale regarding their interest and perceived benefit from the training. An overall score of 35 (sum of all items) on the Likert scale items would be the highest possible score on the measure and would indicate a high level of perceived acceptability of the LGBTQ-affirmative CBT training.
Time Frame: Immediate Post-intervention
Population: This outcome was collected only during the assessment immediately following the intervention for each group.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Immediate Training Group | Waitlist Control Group
Number analyzed (Participants) | 52 | 44
score on a scale | 31.10 (4.17) | 30.57 (5.16)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from baseline through completion of the final follow-up assessment at 8 months.
Arm/Group | Immediate Training Group | Waitlist Control Group
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/60
Other Adverse Events (participants affected / at risk) | 0/61 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT04559698/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/98/NCT04559698/SAP_001.pdf
  • Informed Consent Form (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT04559698/ICF_002.pdf